CLINICAL TRIAL: NCT05826366
Title: Specific Use-results Study of IMJUDO Intravenous Infusion 25mg / IMFINZI Intravenous Infusion 120mg,500mg All Patient Investigation in Patients With Unresectable Advanced or Recurrent Non-small Cell Lung Cancer
Brief Title: Imfinzi/Imjudo NSCLC Japan PMS_Japan Post-Marketing Surveillance (PMS) Study - CEI/SCEI
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D419MC00006
Record Dates: First submitted 2023-04-06; First posted 2023-04-24 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

SUMMARY:
To collect information of safety in patients with unresectable advanced or recurrent non-small cell lung cancer who receive combination therapy of IMJUDO, IMFINZI and other platinum-based anti-cancer agents under actual use in the postmarketing setting.

DETAILED DESCRIPTION:
This investigation will be conducted to collect information of safety in patients with unresectable advanced or recurrent non-small cell lung cancer (NSCLC) who receive combination therapy of IMJUDO Intravenous Infusion 25mg, IMFINZI Intravenous Infusion 120mg, 500mg and other platinum-based anti-cancer agents under actual use in the postmarketing setting.

The investigation will be conducted as one of the additional pharmacovigilance activities in the Japan Risk Management Plan of IMJUDO and IMFINZI in compliance with the Ministerial Ordinance on Good Postmarketing Study Practice (GPSP Ordinance) and for the purpose of application for reexamination under Article 14-4 of the Act on Securing Quality, Efficacy and Safety of Products Including Pharmaceuticals and Medical Devices.

Among the safety specifications defined in the Japan Risk Management Plan of IMJUDO and IMFINZI, the following items are set as the safety specifications for this study.

Interstitial lung disease, Colitis/Severe diarrhoea/Gastrointestinal perforation, Hepatic function disorder/Hepatitis/Cholangitis sclerosing, Endocrine disorders (Dysfunction thyroid, Adrenal dysfunction, Pituitary dysfunction), Type 1 diabetes mellitus, Renal disorder (interstitial nephritis, etc.), Myositis, Myocarditis, Myasthenia gravis, Immune thrombocytopenic purpura, Encephalitis, Severe skin disorder, Nerve disorder (including guillain-barre syndrome), Infusion reaction, Pancreatitis, Rhabdomyolysis, Meningitis, Febrile neutropenia during combination treatment with chemotherapy, Embryo-fetal toxicity, Use in patients with a history of organ transplant (including haematopoietic stem cell transplant)

ELIGIBILITY:
Inclusion Criteria:

* All patients who receive IMJUDO, IMFINZI and other platinum-based anti-cancer agents for their unresectable advanced or recurrent NSCLC

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with unresectable advanced or recurrent NSCLC
Sampling Method: Non-Probability Sample
Enrollment: 296 (Actual)
Dates: Start 2023-06-02 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Incidence of ADRs | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Toshimitsu Tokimoto, Study Director — AstraZeneca KK
Locations (28):
- Japan (28):
  - Research Site, Aichi
  - Research Site, Chiba
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Gifu
  - Research Site, Gunma
  - Research Site, Hiroshima
  - Research Site, Hokkaido
  - Research Site, Hyōgo
  - Research Site, Ibaraki
  - Research Site, Ishikawa
  - Research Site, Kagawa
  - Research Site, Kanagawa
  - Research Site, Kyoto
  - Research Site, Mie
  - Research Site, Miyagi
  - Research Site, Miyazaki
  - Research Site, Nara
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Shizuoka
  - Research Site, Tochigi
  - Research Site, Tokyo
  - Research Site, Tottori
  - Research Site, Toyama
  - Research Site, Wakayama
  - Research Site, Yamagata
  - Research Site, Yamaguchi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home